CLINICAL TRIAL: NCT02446925
Title: Surefire Catheter Versus Standard End-hole Microcatheter in Yttrium-90 Distribution and Tissue Penetration: A Pilot Study
Brief Title: Surefire Catheter Versus Standard End-hole Microcatheter: A Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient number of subjects meeting inclusion criteria
Sponsor: Wright State University (Other)
Collaborators: Surefire Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: Advarra - 42093
Record Dates: First submitted 2015-05-07; First posted 2015-05-18 (Estimated); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surefire® Infusion System (Experimental): Patients randomized to the Surefire® Infusion System treatment arm will undergo Y-90 glass microsphere embolization with a Surefire catheter.
  Interventions: Device: Surefire® Infusion System
- Standard End-hole catheter (Active Comparator): Patients randomized to the standard end-hole catheter treatment arm will undergo Y-90 glass microsphere embolization with a standard end-hole catheter.
  Interventions: Device: Standard End-hole catheter

INTERVENTIONS:
Device: Surefire® Infusion System — Utilization of Surefire® Infusion System for Y-90 glass microsphere embolization
  Arms: Surefire® Infusion System
Device: Standard End-hole catheter — Utilization of Standard End-hole catheter for Y-90 glass microsphere embolization
  Arms: Standard End-hole catheter

SUMMARY:
The Surefire Infusion System is a novel catheter initially developed to prevent reflux of embolic material into non-target vascular territories. Further research has demonstrated improved penetration and distribution of embolic material into treated arterial territories. The purpose of this study is to compare Y-90 glass microsphere distribution and penetration into cancerous tissue within the liver between a standard endhole catheter and the Surefire Infusion System.

DETAILED DESCRIPTION:
Yttrium-90 (Y-90) radioembolization is a minimally invasive trans-arterial treatment for primary and secondary hepatic malignancies that relies on tumor hypervascularity for concentration of radioactive microspheres. The Surefire® Infusion System (SIS) (Westminster, CO) was developed to reduce non-target embolization which can result in morbid complications, especially those involving radioembolic or drug eluting microspheres. Prior to its introduction, radioembolization and other trans-arterial therapies have been performed with standard end-hole catheters. In addition to providing protection against non-target embolization, studies have demonstrated improved penetration of embolic material (tantalum microspheres and Tc-99M labeled MAA) with the use of the SIS when compared to conventional end-hole catheters. To date, no study has demonstrated improved distribution and penetration of yttrium-90 glass microspheres with the use of the Surefire catheter versus a standard end-hole catheter. Y-90 distribution can be evaluated with the use of immediate post-delivery PET/CT imaging as it creates its own pair production and can be imaged in the immediate post delivery period. PET/CT will demonstrate distribution and the dose to tumors can be calculated. The investigators propose a pilot study comparing yttrium-90 tumor distribution and concentration in patients with hepatocellular carcinoma (HCC) with the use of the SIS versus a standard end-hole catheter.

ELIGIBILITY:
Inclusion Criteria:

* Lobar-only treatments
* Patients with biopsy or radiographically proven hepatocellular carcinoma who are not candidates for transplant, surgical resection or ablative therapy
* Patients 18 years of age and older
* Patients who are able to provide written informed consent

Exclusion Criteria:

* Patients with Barcelona-Clinic Liver Cancer (BCLC) Stage C disease,
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≥ 3,
* Patients who are unable to tolerate Y-90,
* Patients with arterial anatomy unsuitable to place Surefire catheter,
* Patients with uncorrectable coagulopathy,
* Patients with platelets less than 50 (uncorrectable),
* Bilirubin >3 mg/dl,
* AST or ALT>5x upper limit of normal,
* Patients who are unable to tolerate angiography,
* Patients with < 3 months to live,
* Patients who meet the standard Y-90 exclusion criteria according to package insert
* Female patients who are pregnant
* Patients under the age of 18
* Patients who are unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Y-90 distribution and concentration as determined by post embolization PET-CT | Up to 12 months
  Y-90 distribution and concentration within targeted hepatocellular carcinoma as determined by post embolization PET-CT.

SECONDARY OUTCOMES:
Secondary outcome (length of duration for arteriogram) | Up to 12 months
  length of duration for arteriogram
Secondary outcome (fluoro time duration) | Up to 12 months
  fluoro time duration
Secondary outcome (number of vessels requiring coiling) | Up to 12 months
  number of vessels requiring coiling
Secondary outcome (tumor response by Response Evaluation Criteria in Solid Tumors) | Up to 12 months
  tumor response by Response Evaluation Criteria in Solid Tumors (m-RECIST criteria)
Secondary outcome- toxicities (per standard labs: Total bilirubin; Aspartate aminotransferase (AST); Alanine aminotransferase (ALT); Albumin; International Normalized Ratio (INR); Creatinine; Alpha Fetoprotein (AFP)) | Up to 12 months
  toxicities (per standard labs: Total bilirubin; Aspartate aminotransferase (AST); Alanine aminotransferase (ALT); Albumin; International Normalized Ratio (INR); Creatinine; Alpha Fetoprotein (AFP))
Secondary outcome (time to progression of tumor) | Up to 12 months
  time to progression of tumor
Secondary outcome (vessel injury) | Up to 12 months
  vessel injury
Secondary outcome (MELD) | Up to 12 months
  Model for End-Stage Liver Disease (MELD)
Secondary outcome (CPS) | Up to 12 months
  Childs-Pugh Score (CPS)
Secondary outcome (non-target embolization) | Up to 12 months
  non-target embolization
Secondary outcome (time to death from first treatment) | Up to 12 months
  time to death from first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Kauffman, MD, Principal Investigator — Wright State University Boonshoft School of Medicine

REFERENCES:
- [Background] Arepally A, Chomas J, Kraitchman D, Hong K. Quantification and reduction of reflux during embolotherapy using an antireflux catheter and tantalum microspheres: ex vivo analysis. J Vasc Interv Radiol. 2013 Apr;24(4):575-80. doi: 10.1016/j.jvir.2012.12.018. Epub 2013 Feb 23. PMID 23462064